CLINICAL TRIAL: NCT06217497
Title: The Effect of Foot Massage Applied to Patients Undergoing Hemodialysis on Sleep Quality and Fatigue Level:Randomized Controlled Study
Brief Title: The Effect of Foot Massage in Patients Undergoing Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Ayşe Şahin, Assistant Professor (Internal Medicine Nursing), Harran University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hemodialysis and Foot Massage
Record Dates: First submitted 2023-06-23; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Nurse-Patient Relations
Keywords: Foot Massage; Hemodialysis; Nursing; Sleep Quality; Fatigue
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: This study was conducted in a randomized controlled design.
Who Masked: Participant
Masking Description: two groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): After the patients in the experimental group were informed verbally and in writing and consented to participate in the study, the Patient Information Form, the Piper Fatigue Scale (PFS), and the Pittsburgh Sleep Quality Index (PSQI) were applied in the first interview and the initial readings were obtained. The researcher received training on a classical massage from an expert massage therapist before the foot massaging application. Patients in the experimental group were subjected to a foot massage with baby oil for 10 minutes during HD treatment three times a week for four weeks, 12 times in total. At the end of the second and fourth weeks after the foot massage, the second and third readings were recorded by repeating the PFS and PSQI.
  Interventions: Other: Foot massage
- Control Group (No Intervention): Patients in the control group were not subjected to any intervention other than routine HD treatment and nursing care. The first readings were obtained by applying the Patient Information Form, PFS and PSQI at the first interview, and the second and third measurement values were obtained by repeating the PFS and PSQI at the end of the second and fourth weeks.

INTERVENTIONS:
Other: Foot massage — Patients in the experimental group were subjected to a foot massage with baby oil for 10 minutes during HD treatment three times a week for four weeks, 12 times in total. At the end of the second and fourth weeks after the foot massage, the second and third readings were recorded by repeating the PFS and PSQI
  Arms: Experimental Group

SUMMARY:
Hemodialysis patients were divided into experimental and control groups. Foot massage was applied to the patients in the experimental group. Foot massage was not applied to the patients in the control group and routine nursing care was provided. Pre-test, mid-test and post-test sleep quality and fatigue level scores of the patients were determined.

DETAILED DESCRIPTION:
An experimental study design was used to conduct this research on 73 hemodialysis patients treated in a hemodialysis unit. The aim of this study is to investigate how foot massage applied to hemodialysis patients affects sleep quality and fatigue level.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria were determined as follows:

  * Having a PSQI score of 5 points and above
  * Receiving HD treatment for at least 6 months
  * Having no neuropathy d) Using no sleeping pills
  * Having no communication problem
  * Having full orientation and no psychiatric problems
  * Having no conditions in the lower extremities and feet that would preclude massaging (no open wounds on the skin, orthopaedic and joint problems, oedema, abscess, infection, thrombophlebitis, deep vein thrombosis, thrombocytopenia, etc.)
  * Having no history of allergy to the oil used for massage.

Exclusion Criteria:

Exclusion criteria were determined as follows:

* Receiving less than 6 months of HD treatment
* Having communication problem
* Suffering from neuropathy
* Having incomplete orientation and any psychiatric problem
* Having a PSQI score below 5
* Having conditions in the lower extremities and feet that would preclude massaging (open wounds on the skin, orthopaedic and joint problems, oedema, abscess, infection, thrombophlebitis, deep vein thrombosis, thrombocytopenia, etc.) and having a history of allergy to the oil used for massage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Piper fatigue scale | Last 2 weeks and last 4 weeks
  Piper Fatigue Scale (PFS) was developed by Piper et al. The scale consists of a total of 22 items. Each item is rated over 0-10 points through Visual Analogue Scale (VAS) under four subscales related to the patient's subjective perception of fatigue. The behavioural subscale consists of 6 items (2-7), the affective subscale consists of 5 items (8-12), the sensory subscale consists of 5 items (13-17), and the cognitive subscale consists of 6 items [18-23]. Total fatigue score and subscale scores are calculated over 22 items. Items 1, 24, 25, 26 and 27 in the scale are not used in calculating the fatigue score. Total fatigue score is obtained by summing the items and dividing the resultant value by the total number of items, and subscale scores are obtained by summing the scores of all items in that subscale and dividing the resultant value by the number4 of items.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | Last 2 weeks and last 4 weeks
  The Pittsburgh Sleep Quality Index (PSQI) was developed by Buysse et al., . Turkish validity and reliability study of the scale was conducted by Ağargün et al.,. The index, which evaluates sleep quality, sleep duration, sleep latency, sleep disturbance and severity in the last 4 weeks, consists of a total of 24 items. 19 items in the index are self-assessment questions, the last 5 questions are answered by the individual's roommate or spouse, and the last 5 questions are not included in the scoring. There are seven components of the PSQI (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping medication, daytime dysfunction). The sum of these seven components gives the total PSQI score. Total score ranges from 0-21, and each item gets a score between 0-3 points. A PSQI total score of 5 points and above indicates that the sleep quality is "poor" and a higher score indicates more sleep complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan Çıtlık SARITAŞ, PhD, Principal Investigator — Turgut ÖZAL University
Locations (1):
- Harran University, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study was conducted in a randomized controlled manner with experimental and control groups.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: No time limit
Access Criteria: All data
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp